CLINICAL TRIAL: NCT01186770
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Study of Oral Methylnaltrexone for the Treatment of Opioid-Induced Constipation in Subjects With Chronic, Non-Malignant Pain
Brief Title: A Study of Oral Methylnaltrexone (MNTX) for the Treatment of Opioid-Induced Constipation (OIC) in Participants With Chronic, Non-Malignant Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MNTX 3201
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Opioid-Induced Constipation
Keywords: Treatment of Opioid-Induced Constipation in Participants with Chronic, Non-Malignant Pain
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MNTX 150 mg (Experimental): Participants will receive methylnaltrexone (MNTX) 150 milligrams (mg) (1 tablet of MNTX 150 mg and 2 matching placebo tablets) orally once daily (QD) for 28 days (4 weeks), then MNTX tablets at a dose as needed (PRN) for remaining 56 days (8 weeks).
  Interventions: Drug: Methylnaltrexone; Drug: Placebo
- MNTX 300 mg (Experimental): Participants will receive MNTX 300 mg (2 tablets of MNTX 150 mg each and 1 matching placebo tablet) orally QD for 28 days (4 weeks), then MNTX tablets at a dose PRN for remaining 56 days (8 weeks).
  Interventions: Drug: Methylnaltrexone; Drug: Placebo
- MNTX 450 mg (Experimental): Participants will receive MNTX 450 mg (3 tablets of MNTX 150 mg each) orally QD for 28 days (4 weeks), then MNTX tablets at a dose PRN for remaining 56 days (8 weeks).
  Interventions: Drug: Methylnaltrexone
- Placebo (Placebo Comparator): Participants will receive 3 tablets of placebo matched to MNTX orally QD for 84 days (12 weeks).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone — Methylnaltrexone will be administered as per the dose and schedule specified in the respective arms.
  Other Names: Relistor
  Arms: MNTX 150 mg; MNTX 300 mg; MNTX 450 mg
Drug: Placebo — Placebo matching to methylnaltrexone will be administered as per the schedule specified in the respective arms.
  Arms: MNTX 150 mg; MNTX 300 mg; Placebo

SUMMARY:
MNTX 3201 is a Phase 3, international, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the safety and efficacy of oral MNTX for the treatment of opioid induced constipation in participants with chronic, non-malignant pain.

ELIGIBILITY:
Key Inclusion Criteria:

1. History of chronic non-malignant pain (originating from a non-malignant source) with condition(s) underlying the chronic pain of greater than or equal to (≥) 2 months' duration before the screening visit.
2. Taking oral, transdermal, intravenous (IV), or subcutaneous (SC) opioids for chronic non-malignant pain for ≥1 month.
3. No known history of chronic constipation prior to the initiation of opioid therapy.
4. Currently taking laxative therapy for ≥30 days and willing to discontinue all laxative therapy at the start of screening period and use only study-permitted rescue laxatives throughout the screening and double-blind treatment periods..

Key Exclusion Criteria:

1. Prior treatment with oral MNTX.
2. Prior treatment with SC MNTX within 30 days of screening.
3. Women who are pregnant, breastfeeding, or plan to become pregnant during the study.
4. Fecal incontinence, rectal prolapse, fecal ostomy or other clinically significant gastrointestinal disorders such as inflammatory bowel disease or clinically significant irritable bowel syndrome that would have made bowel movement assessment inaccurate.
5. Current treatment with partial opioid agonists (for example; buprenorphine) or combination agonists/antagonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 804 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2011-09-08 (Actual); Study Completion 2011-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (2):
- United States (2):
  - PRA International, Raleigh, North Carolina
  - PRA, Intl., Raleigh, North Carolina

REFERENCES:
- [Derived] Liao SS, Slatkin NE, Stambler N. The Influence of Age on Central Effects of Methylnaltrexone in Patients with Opioid-Induced Constipation. Drugs Aging. 2021 Jun;38(6):503-511. doi: 10.1007/s40266-021-00850-w. Epub 2021 Mar 31. PMID 33788162

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 804 participants met inclusion/exclusion criteria and randomized in 1:1:1:1 ratio to either MNTX 150 mg, MNTX 300 mg, MNTX 450 mg, or placebo treatment groups.
Groups:
- MNTX 150 mg: Participants received methylnaltrexone (MNTX) 150 milligrams (mg) (1 tablet of MNTX 150 mg and 2 matching placebo tablets) orally once daily (QD) for 28 days (4 weeks), then MNTX tablets at a dose as needed (PRN) for remaining 56 days (8 weeks).
- MNTX 300 mg: Participants received MNTX 300 mg (2 tablets of MNTX 150 mg each and 1 matching placebo tablet) orally QD for 28 days (4 weeks), then MNTX tablets at a dose PRN for remaining 56 days (8 weeks).
- MNTX 450 mg: Participants received MNTX 450 mg (3 tablets of MNTX 150 mg each) orally QD for 28 days (4 weeks), then MNTX tablets at a dose PRN for remaining 56 days (8 weeks).
- Placebo: Participants received 3 tablets of placebo matched to MNTX orally QD for 84 days (12 weeks).
Period: Overall Study
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo
Started | 201 | 202 | 200 | 201
Intent-to-treat (ITT Population) (Received at least 1 dose of study drug) | 201 | 201 | 200 | 201
Completed | 160 | 156 | 148 | 143
Not Completed | 41 | 46 | 52 | 58
Not completed — Ineligibility | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 7 | 9 | 12 | 14
Not completed — Adverse Event | 2 | 9 | 7 | 9
Not completed — Withdrawal by Subject | 15 | 13 | 11 | 17
Not completed — Lost to Follow-up | 10 | 6 | 14 | 9
Not completed — Insufficient response to treatment | 7 | 8 | 5 | 7
Not completed — Other than specified | 0 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Groups:
- MNTX 150 mg: Participants received MNTX 150 mg (1 tablet of MNTX 150 mg and 2 matching placebo tablets) orally QD for 28 days (4 weeks), then MNTX tablets at a dose PRN for remaining 56 days (8 weeks).
- Total: Total of all reporting groups
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo | Total
Number analyzed (Participants) | 201 | 201 | 200 | 201 | 803
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 0 | 0 | 1
  Between 18 and 65 years | 185 | 182 | 181 | 179 | 727
  >=65 years | 15 | 19 | 19 | 22 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (10.32) | 51.5 (10.54) | 51.4 (10.50) | 52.6 (10.33) | 51.6 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 114 | 128 | 130 | 505
  Male | 68 | 87 | 72 | 71 | 298
Primary pain condition requiring opioid medication [Count of Participants; unit: Participants]
  Back pain | 132 | 136 | 135 | 145 | 548
  Joint/extremity pain | 13 | 16 | 11 | 10 | 50
  Arthritis | 20 | 15 | 19 | 12 | 66
  Neurologic/neuropathic pain | 16 | 13 | 16 | 11 | 56
  Fibromyalgia | 15 | 8 | 11 | 12 | 46
  Other pain condition requiring opioids | 5 | 13 | 8 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Average Percentage of Dosing Days That Resulted in Rescue-Free Bowel Movements (RFBMs) Within 4 Hours of Dosing During Weeks 1 to 4
Description: RFBM was defined as a bowel movement without laxative use within 24 hours prior to bowel movement.
Time Frame: Weeks 1 to 4
Population: ITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo
Number analyzed (Participants) | 201 | 201 | 200 | 201
percentage of days | 21.05 (20.116) | 24.64 (21.311) | 27.40 (23.453) | 18.18 (16.995)
Statistical Analysis 1: Comparison: MNTX 150 mg vs Placebo; Analysis was performed using analysis of covariance (ANCOVA) with treatment as effect and analysis region as covariate; Test type: Superiority; p = 0.1692, ANCOVA — Threshold for significance at 0.0167 level; Least square (LS) mean difference = 2.83, 95% CI [-1.21 to 6.86]
Statistical Analysis 2: Comparison: MNTX 300 mg vs Placebo; Analysis was performed using ANCOVA with treatment as effect and analysis region as covariate; Test type: Superiority; p = 0.0016, ANCOVA — Threshold for significance at 0.0167 level; LS mean difference = 6.51, 95% CI 2-sided [2.47 to 10.55]
Statistical Analysis 3: Comparison: MNTX 450 mg vs Placebo; Analysis was performed using ANCOVA with treatment as effect and analysis region as covariate; Test type: Superiority; p < 0.0001, ANCOVA — Threshold for significance at 0.0167 level; LS mean difference = 9.13, 95% CI 2-sided [5.09 to 13.18]

2. Secondary Outcome: Percentage of Participants Who Responded (Responder) to Study Drug During Weeks 1 to 4
Description: A responder was defined as at least 3 RFBMs/week, with an increase of at least 1 RFBM/week over baseline, for at least 3 out of the first 4 weeks of the treatment period. Weekly number of RFBMs were calculated as follows: 7 * total number of RFBMs in a week/all non-missing assessment days in the given week. Weekly number of RFBMs was set to missing for any week when a participant completed less than (<) 4 diary days in a week. A RFBM was a bowel movement without laxative use within 24 hrs prior to the bowel movement.
Time Frame: Weeks 1 to 4
Population: ITT population included all randomized participants who received at least 1 dose of study drug. Missing data was imputed using last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo
Number analyzed (Participants) | 201 | 201 | 200 | 201
percentage of participants | 45.3 | 51.7 | 54.5 | 40.8
Statistical Analysis 1: Comparison: MNTX 150 mg vs Placebo; Analysis was performed using logistic regression model with treatment as effect and analysis region as covariate; Test type: Superiority; p = 0.3076, Regression, Logistic — Threshold for significance at 0.0167 level; Odds Ratio (OR) = 1.23, 95% CI 2-sided [0.82 to 1.84]
Statistical Analysis 2: Comparison: MNTX 300 mg vs Placebo; Analysis was performed using logistic regression model with treatment as effect and analysis region as covariate; Test type: Superiority; p = 0.0339, Regression, Logistic — Threshold for significance at 0.0167 level; Odds Ratio (OR) = 1.54, 95% CI 2-sided [1.03 to 2.29]
Statistical Analysis 3: Comparison: MNTX 450 mg vs Placebo; Analysis was performed using logistic regression model with treatment as effect and analysis region as covariate; Test type: Superiority; p = 0.0043, Regression, Logistic — Threshold for significance at 0.0167 level; Odds Ratio (OR) = 1.79, 95% CI [1.20 to 2.66]

3. Secondary Outcome: Change in Weekly Number of RFBMs From Baseline Over the Entire First 4 Weeks (28 Days) of Dosing
Description: Weekly number of RFBMs were calculated as follows: 7 * total number of RFBMs in a week/all non-missing assessment days in the given week. Weekly number of RFBMs was set to missing for any week when a participant completed less than (<) 4 diary days in a week. A RFBM was a bowel movement without laxative use within 24 hrs prior to the bowel movement.
Time Frame: Baseline, Weeks 1 to 4
Population: ITT population included all randomized participants who received at least 1 dose of study drug. Missing data was imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: RFBMs
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo
Number analyzed (Participants) | 201 | 201 | 200 | 201
RFBMs
  Baseline | 1.46 (0.911) | 1.35 (0.891) | 1.37 (0.789) | 1.49 (1.045)
  Change during Weeks 1-4 | 1.98 (2.139) | 2.43 (2.616) | 2.44 (2.515) | 1.87 (2.052)
Statistical Analysis 1: Comparison: MNTX 150 mg vs Placebo; Analysis was performed using ANCOVA model with treatment as effect and analysis region and baseline as covariates; Test type: Superiority; p = 0.6920, ANCOVA — Threshold for significance at 0.0167 level; LS mean difference = 0.09, 95% CI 2-sided [-0.36 to 0.55]
Statistical Analysis 2: Comparison: MNTX 300 mg vs Placebo; Analysis was performed using ANCOVA model with treatment as effect and analysis region and baseline as covariates; Test type: Superiority; p = 0.0274, ANCOVA — Threshold for significance at 0.0167 level; LS mean difference = 0.51, 95% CI 2-sided [0.06 to 0.97]
Statistical Analysis 3: Comparison: MNTX 450 mg vs Placebo; Analysis was performed using ANCOVA model with treatment as effect and analysis region and baseline as covariates; Test type: Superiority; p = 0.0237, ANCOVA — Threshold for significance at 0.0167 level; LS mean difference = 0.53, 95% CI 2-sided [0.07 to 0.98]

ADVERSE EVENTS:
Time Frame: Baseline (Day 1) up to Day 98
Description: Adverse events were collected by non-systematic (participant reports) and systematic methods (investigator examinations and lab tests). For both adverse events tables, a participant reporting more than one adverse event for a particular MedDRA preferred term or system organ class was counted only once for that MedDRA preferred term or system organ class.
Arm/Group | MNTX 150 mg | MNTX 300 mg | MNTX 450 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/201 | 6/201 | 4/200 | 8/201
Other Adverse Events (participants affected / at risk) | 38/201 | 35/201 | 42/200 | 32/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MNTX 150 mg (N=201) | MNTX 300 mg (N=201) | MNTX 450 mg (N=200) | Placebo (N=201)
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myositis ossificans (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 | 0
Spinal fusion surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MNTX 150 mg (N=201) | MNTX 300 mg (N=201) | MNTX 450 mg (N=200) | Placebo (N=201)
Abdominal pain (Gastrointestinal disorders) | 11 | 16 | 21 | 17
Diarrhoea (Gastrointestinal disorders) | 7 | 13 | 16 | 7
Flatulence (Gastrointestinal disorders) | 11 | 7 | 10 | 9
Nausea (Gastrointestinal disorders) | 13 | 16 | 12 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 6 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.